CLINICAL TRIAL: NCT06271850
Title: Effect of Pilates Exercises on Forward Head Posture in Breastfeeding Women: A Randomized Controlled Trial
Brief Title: Effect of Pilates Exercises on Forward Head Posture in Breastfeeding Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Onsy Ewass, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004949
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-02

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ergonomic breastfeeding training (control group) (Active Comparator): They will receive ergonomics breastfeeding training only.
  Interventions: Other: Ergonomics breastfeeding training
- Pilates exercises and ergonomic breastfeeding training (study group) (Experimental): They will receive Pilates exercises, in addition to ergonomics breastfeeding training.
  Interventions: Other: Ergonomics breastfeeding training; Other: Pilates exercises

INTERVENTIONS:
Other: Ergonomics breastfeeding training — The ergonomics training includes the most ergonomically appropriate methods to breastfeed and ergonomic guidelines, including how to cuddle and breastfeed the baby correctly.
Other: Pilates exercises — Pilates exercises, 3 times per week, for 8 weeks, in the form of neck extensor stretching, neck extensor and rotation stretching, pectoral muscle stretching, strengthening of deep neck flexors and scapular retractor, and core strengthening exercises ( pelvic bridging, plank, cat and camel, curl up, single leg abdominal press and double leg abdominal press).
  Arms: Pilates exercises and ergonomic breastfeeding training (study group)

SUMMARY:
Musculoskeletal postural issues stemming from infant care positions can exert a significant impact on the cervical, thoracic, and lumbar spine. These positions can induce mechanical alterations in the spine's natural curvature, potentially resulting in long-term deformities in postnatal women such as forward head posture (FHP), ultimately contributing to physical disability over the long term.so, The purpose of this study is to determine the effect of Pilates exercises on FHP in breastfeeding women.

DETAILED DESCRIPTION:
seventy-four breastfeeding women having forward head posture (FHP) will participate in this study. They will be selected randomly from the outpatient clinic of orthopedic of Suez Canal Authority Hospital in Portsaid, Egypt.

Group (A) (Control group): will consist of 37 breastfeeding women. They will receive ergonomic breastfeeding training for 8 weeks.

Group (B) (Study group): will consist of 37 breastfeeding women. They will receive the same ergonomic breastfeeding training plus Pilates exercises 3 times per week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* All women are breastfeeding and will have FHP.
* They are between six to twelve months post-delivery.
* They should have a single, healthy, and full-term baby without complications.
* Their body mass index (BMI) will not exceed 30 Kg/m2.
* Their parity will range from 2 to 3 children.
* They are housewife.

Exclusion Criteria:

* Cancer of the breast or the surrounding area, any previous breast or chest surgery, breast infection, retracted, cracked, inflamed or inverted nipples.
* Any cardiorespiratory disease, anemia, or diabetes mellitus.
* Recent fracture or surgery of the cervical spine or shoulder.
* History of physical and mental diseases.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-20 (Actual)

PRIMARY OUTCOMES:
Measurement of craniovertebral angle (CVA) | up to 8 weeks
  It will be measured before and after treatment program by using posture screen analysis mobile application. This method has many advantages, as it is relatively fast, the image and values obtained are easily preserved, and it is more precise and reliable than visual evaluation alone The CVA is the best indicator of FHP. To determine this angle, two references are defined: One line that runs from the swallow of the ear to seventh cervical vertebra (C7) and another horizontal line parallel to the ground that passes only through the spinous apophysis of C7. An angle of less than 50°-53° may indicate FHP. Thereby, the smaller the CVA, the greater the disability
Assessment of neck pain intensity | up to 8 weeks
  It will be evaluated before and after treatment program by using VAS, which is a linear scale that measures the magnitude of pain severity. It encompasses a horizontal line scaled as a spectrum from mild pain beginning from the left to increasing severity to the right end of the horizontal line. The line is 10 cm in length, with each side of the line ending in extremes either no pain or intense pain. In terms of utilization, each participant will mark her pain on the line of the spectrum of the scale
Measurement of cervical range of motion | up to 8 weeks
  It will be measured before and after treatment program by goniometer. The movements that will measured by the goniometer include flexion and extension, right and left lateral flexion, and right and left rotation. The goniometer will be placed on the participant's head. During all the measurements, the participant will be seated, with her back straight, and looking ahead; her feet will be supported on the floor. The participant will remain in the same sitting position from the moment the recording procedure will start. The measurement will be performed from "the neutral" position to the final range of motion in a given plane. The participant will perform a practice trial. During each trial, the movement will be executed to reflect the participant's maximum capabilities. When the maximum movement will be performed in one direction, the final position will be identified and recorded

SECONDARY OUTCOMES:
Evaluation of disability due to neck pain | up to 8 weeks
  It will be evaluated before and after treatment program by the neck disability index, which is a well-validated 10-item questionnaire, with each item rated on a 0 to 5-point scale. The sum of the 10 items gives a score between 0-50. The lower the score, the less self-rated the disability. 0-4 = no disability, 5-14 = mild disability, 15-24 = moderate disability, 25-34 = severe disability, 35 or over = complete disability
Assessment of neck muscle fatigue | up to 8 weeks
  It will be assessed before and after treatment program by the FSS questionnaire, which contains nine statements that rate the severity of fatigue symptoms. The participant will read each statement and circle a number from 1 to 7, based on how accurately it reflects her condition A low value indicates strong disagreement with the statement, whereas a high value indicates strong agreement. A total score of less than 36 suggests that participant may not be suffering from fatigue. A total score of 36 or more suggests that participant may be suffering from fatigue.
Assessment of breastfeeding self-efficacy | up to 8 weeks
  It will be measured before and after treatment program by using Breastfeeding Self Efficacy Scale Short Form (BSES-SF), which represents a 14-item self-administered instrument derived from the original 33-item BSES that measures breastfeeding confidence. All items are preceded by the phrase ''I can always'' and rated on a 5-point Likert scale, ranging from 1 (not at all confident) to 5 (always confident). Total scores range from 14 to 70, with higher scores reflecting more significant levels of breastfeeding self-efficacy.
Measurement of weight and height of baby | up to 8 weeks
  It will be assessed before and after treatment program by using a weighing scale and a length board. The weighing scale will be calibrated then each baby in both groups will be placed over the scale wearing only the under wears and without the baby diapers two times and the average of the two readings will be taken. Each baby's length will be measured in a recumbent position using a length board which should be placed on a flat, stable surface such as a table.
Assessment of Health-Related Quality of Life | up to 8 weeks
  It will be assessed before and after treatment program using Free online 36- item short form health survey (SF-36) score calculator. It measures eight scales: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Component analyses showed that there are two distinct concepts measured by the SF-36: a physical dimension, represented by the Physical Component Summary (PCS), and a mental dimension, represented by the Mental Component Summary (MCS). its value ranges from 0-100. 0 indicates the worst health state and 100 indicates the best health state.

CONTACTS AND LOCATIONS:
Overall Officials: Khadega S Abd El Aziz, PHD, Study Chair — Cairo University
Locations (1):
- Doaa Onsy Ewass, Port Said, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF